CLINICAL TRIAL: NCT03098667
Title: Study of the Laryngopharyngeal Symptoms After Minimally Invasive Thyroidectomy: Comparison Between the Protector Laryngeal Mask Airway and the Endotracheal Tube.
Brief Title: Laryngeal Mask Airway (LMA) Protector for Minimally Invasive Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 424 General Military Hospital (Other)
Responsible Party: Principal Investigator, Georgios Kotsovolis, Dr Georgios Kotsovolis, 424 General Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 184/15.03.2017
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Sore Throat; Dysphagia; Postoperative Pain
MeSH Terms: conditions — Pharyngitis; Deglutition Disorders; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LMA Protector (Experimental): After induction of general anesthesia, the LMA Protector will be applied for airway management. The size of the laryngeal mask will be chosen according to the manufacturer's instructions. Lubricant gel will be applied to the dorsal side of the mask to ease the insertion to the oropharynx. The cuff of the mask will be filled with air by syringe until the indication of the integrated cuff pressure indicator is appropriate according to the manufacturer (green indication). If the indication changes during surgery, air will be added or removed accordingly. If the ventilation of the patient is inadequate at the beginning or anytime during the operation, the mask will be removed and the patient will be intubated
  Interventions: Device: LMA Protector
- Endotracheal tube (Active Comparator): After induction of general anesthesia, the endotracheal tube be applied for airway management. The size of the tube will be 7.5 for female and 8.5 for male patients. The cuff of of the tube will be filled with 10ml air.
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: LMA Protector — After induction of general anesthesia, the LMA Protector will be applied for airway management. The size of the laryngeal mask will be chosen according to the manufacturer's instructions. Lubricant gel will be applied to the dorsal side of the mask to ease the insertion to the oropharynx. The cuff of the mask will be filled with air by syringe until the indication of the integrated cuff pressure indicator is appropriate according to the manufacturer (green indication). If the indication changes during surgery, air will be added or removed accordingly. If the ventilation of the patient is inadequate at the beginning or anytime during the operation, the mask will be removed and the patient will be intubated.
  Arms: LMA Protector
Device: Endotracheal tube — After induction of general anesthesia, the endotracheal tube be applied for airway management. The size of the tube will be 7.5 for female and 8.5 for male patients. The cuff of of the tube will be filled with 10ml air.
  Arms: Endotracheal tube

SUMMARY:
The patients will be allocated to 2 groups: the LMA group and the endotracheal tube (ET) group. Airway management will be done with the LMA Protector for the patients of the LMA group and with the classic endotracheal tube for the patients of the ET group. The main purpose of the study is to determine if the application of the LMA Protector causes less laryngopharyngeal symptoms than the endotracheal tube after minimally invasive thyroidectomy. The secondary purpose is to confirm that the LMA Protector is a safe alternative airway management device for minimally invasive thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Total thyroidectomy with the minimally invasive method.
* American Society of Anesthesiologists (ASA) classification 1-3

Exclusion Criteria:

* Clinical conditions which cause any kind of airway obstruction or compromise.
* Tracheal displacement greater than 2cm from midline.
* History of gastroesophageal reflux disease.
* Expected difficult airway.
* History of impossible intubation.
* BMI>35
* Reoperation within 24hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Postoperative sore throat. | Within 20 minutes from the end of the procedure.
  The patients will be asked to evaluate their postoperative constant pharyngeal pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative sore throat. | 1 hour after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative constant pharyngeal pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative sore throat. | 6 hours after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative constant pharyngeal pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative sore throat. | 12 hours after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative constant pharyngeal pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative sore throat. | 24 hours after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative constant pharyngeal pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative surgical site pain. | Within 20 minutes from the end of the procedure.
  The patients will be asked to evaluate their postoperative surgical trauma pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative surgical site pain. | 1 hour after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative surgical trauma pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative surgical site pain. | 6 hours after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative surgical trauma pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative surgical site pain. | 12 hours after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative surgical trauma pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative surgical site pain. | 24 hours after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative surgical trauma pain by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative dysphagia. | Within 20 minutes from the end of the procedure.
  The patients will be asked to evaluate their postoperative pharyngeal pain caused after swallowing one sip of water by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative dysphagia. | 1 hour after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative pharyngeal pain caused after swallowing one sip of water by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative dysphagia. | 6 hours after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative pharyngeal pain caused after swallowing one sip of water by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative dysphagia. | 12 hours after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative pharyngeal pain caused after swallowing one sip of water by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).
Postoperative dysphagia. | 24 hours after the exit from the recovery room.
  The patients will be asked to evaluate their postoperative pharyngeal pain caused after swallowing one sip of water by using the 11grade Numerical Rating Scale (0 no pain, 10 maximum possible pain).

SECONDARY OUTCOMES:
Airway management difficulty. | 3 minutes after induction of general anesthesia.
  The efforts required to establish a secure airway and manage adequate patient ventilation will be recorded.
Airway management complications. | Within 5 minutes from induction of general anesthesia.
  Any complication from airway management will be recorded like bleeding from the stomatopharynx or the larynx, tooth trauma, lip trauma, etc.
Emergence coughing. | Within 10 minutes from the end of the surgery.
  The incidence of cough upon emergence from general anesthesia will be recorded.
Postoperative paracetamol consumption. | 1, 6, 12 and 24 hours after emergence from general anesthesia.
  The patients will be instructed to ask for analgesics as needed. When rescue analgesia is required 1000mg paracetamol will be administered. The frequency of paracetamol administration will be documented.
Postoperative hoarseness. | Within 20 minutes from the end of the procedure and after 1, 6, 12 and 24 hours.
  The patients postoperative hoarseness will be evaluated according to the GRBAS scale.

CONTACTS AND LOCATIONS:
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chun BJ, Bae JS, Lee SH, Joo J, Kim ES, Sun DI. A prospective randomized controlled trial of the laryngeal mask airway versus the endotracheal intubation in the thyroid surgery: evaluation of postoperative voice, and laryngopharyngeal symptom. World J Surg. 2015 Jul;39(7):1713-20. doi: 10.1007/s00268-015-2995-7. PMID 25670039
- [Background] Kumar C, Mishra A. Prospective randomized controlled trial on the use of flexible reinforced laryngeal mask airway (LMA) during total thyroidectomy: effects on postoperative laryngopharyngeal symptoms: reply. World J Surg. 2015 Mar;39(3):810. doi: 10.1007/s00268-014-2675-z. No abstract available. PMID 24981369
- [Background] Moris D, Mantonakis E, Makris M, Michalinos A, Vernadakis S. Hoarseness after thyroidectomy: blame the endocrine surgeon alone? Hormones (Athens). 2014 Jan-Mar;13(1):5-15. doi: 10.1007/BF03401316. PMID 24722123
- [Background] Ryu JH, Yom CK, Park DJ, Kim KH, Do SH, Yoo SH, Oh AY. Prospective randomized controlled trial on the use of flexible reinforced laryngeal mask airway (LMA) during total thyroidectomy: effects on postoperative laryngopharyngeal symptoms. World J Surg. 2014 Feb;38(2):378-84. doi: 10.1007/s00268-013-2269-1. PMID 24146195
- [Background] Nemr K, Simoes-Zenari M, Cordeiro GF, Tsuji D, Ogawa AI, Ubrig MT, Menezes MH. GRBAS and Cape-V scales: high reliability and consensus when applied at different times. J Voice. 2012 Nov;26(6):812.e17-22. doi: 10.1016/j.jvoice.2012.03.005. Epub 2012 Sep 29. PMID 23026732
- [Background] Taguchi A, Mise K, Nishikubo K, Hyodo M, Shiromoto O. Japanese version of voice handicap index for subjective evaluation of voice disorder. J Voice. 2012 Sep;26(5):668.e15-9. doi: 10.1016/j.jvoice.2011.11.005. Epub 2012 Jan 30. PMID 22285453
- [Background] Awan SN, Helou LB, Stojadinovic A, Solomon NP. Tracking voice change after thyroidectomy: application of spectral/cepstral analyses. Clin Linguist Phon. 2011 Apr;25(4):302-20. doi: 10.3109/02699206.2010.535646. Epub 2010 Dec 15. PMID 21158501
- [Background] Werth K, Voigt D, Dollinger M, Eysholdt U, Lohscheller J. Clinical value of acoustic voice measures: a retrospective study. Eur Arch Otorhinolaryngol. 2010 Aug;267(8):1261-71. doi: 10.1007/s00405-010-1214-2. Epub 2010 Feb 21. PMID 20567980
- [Background] Maryn Y, De Bodt M, Roy N. The Acoustic Voice Quality Index: toward improved treatment outcomes assessment in voice disorders. J Commun Disord. 2010 May-Jun;43(3):161-74. doi: 10.1016/j.jcomdis.2009.12.004. Epub 2009 Dec 23. PMID 20080243
- [Background] Pott L, Swick JT, Stack BC Jr. Assessment of recurrent laryngeal nerve during thyroid surgery with laryngeal mask airway. Arch Otolaryngol Head Neck Surg. 2007 Mar;133(3):266-9. doi: 10.1001/archotol.133.3.266. PMID 17372084
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Brimacombe J, Knott J, Keller C. Laryngeal mask airway for preservation of the external branch of the superior laryngeal nerve during thyroid surgery. Can J Anaesth. 2003 Oct;50(8):858. doi: 10.1007/BF03019391. No abstract available. PMID 14525838
- [Background] Scheuller MC, Ellison D. Laryngeal mask anesthesia with intraoperative laryngoscopy for identification of the recurrent laryngeal nerve during thyroidectomy. Laryngoscope. 2002 Sep;112(9):1594-7. doi: 10.1097/00005537-200209000-00011. PMID 12352669
- [Background] Rosswick P. Use of the laryngeal mask airway in thyroid and parathyroid surgery as an aid in identification and preservation of the recurrent laryngeal nerves. Ann R Coll Surg Engl. 2002 Mar;84(2):148; author reply 148. No abstract available. PMID 11995766
- [Background] Watters G. Use of the laryngeal mask airway in thyroid and parathyroid surgery as an aid in identification and preservation of the recurrent laryngeal nerves. Ann R Coll Surg Engl. 2002 Mar;84(2):148; author reply 148. No abstract available. PMID 11995765
- [Background] Dingle AF. Use of the laryngeal mask airway in thyroid and parathyroid surgery as an aid in identification and preservation of the recurrent laryngeal nerves. Ann R Coll Surg Engl. 2002 Mar;84(2):147; author reply 148. No abstract available. PMID 11995764
- [Background] Shah EF, Allen JG, Greatorex RA. Use of the laryngeal mask airway in thyroid and parathyroid surgery as an aid to the identification and preservation of the recurrent laryngeal nerves. Ann R Coll Surg Engl. 2001 Sep;83(5):315-8. PMID 11806554
- [Background] Palazzo FF, Allen JG, Greatorex RA. Laryngeal mask airway and fibre-optic tracheal inspection in thyroid surgery: a method for timely identification of tracheomalacia requiring tracheostomy. Ann R Coll Surg Engl. 2000 Mar;82(2):141-2. PMID 10743437
- [Background] Wuyts FL, De Bodt MS, Van de Heyning PH. Is the reliability of a visual analog scale higher than an ordinal scale? An experiment with the GRBAS scale for the perceptual evaluation of dysphonia. J Voice. 1999 Dec;13(4):508-17. doi: 10.1016/s0892-1997(99)80006-x. PMID 10622517
- [Background] Rieger A, Brunne B, Striebel HW. Intracuff pressures do not predict laryngopharyngeal discomfort after use of the laryngeal mask airway. Anesthesiology. 1997 Jul;87(1):63-7. doi: 10.1097/00000542-199707000-00009. PMID 9232135
- [Background] Rieger A, Brunne B, Hass I, Brummer G, Spies C, Striebel HW, Eyrich K. Laryngo-pharyngeal complaints following laryngeal mask airway and endotracheal intubation. J Clin Anesth. 1997 Feb;9(1):42-7. doi: 10.1016/S0952-8180(96)00209-7. PMID 9051545
- [Background] Hobbiger HE, Allen JG, Greatorex RG, Denny NM. The laryngeal mask airway for thyroid and parathyroid surgery. Anaesthesia. 1996 Oct;51(10):972-4. doi: 10.1111/j.1365-2044.1996.tb14969.x. PMID 8984876
- [Background] Premachandra DJ. Application of the laryngeal mask airway to thyroid surgery and the preservation of the recurrent laryngeal nerve. Ann R Coll Surg Engl. 1992 May;74(3):226. No abstract available. PMID 1616271
- [Background] Charters P, Cave-Bigley D. Application of the laryngeal mask airway to thyroid surgery and the preservation of the recurrent laryngeal nerve. Ann R Coll Surg Engl. 1992 May;74(3):225-6. No abstract available. PMID 1616270
- [Background] Maroof M, Siddique M, Khan RM. Post-thyroidectomy vocal cord examination by fibreoscopy aided by the laryngeal mask airway. Anaesthesia. 1992 May;47(5):445. doi: 10.1111/j.1365-2044.1992.tb02238.x. No abstract available. PMID 1599080
- [Background] Charters P, Cave-Bigley D, Roysam CS. Should a laryngeal mask be routinely used in patients undergoing thyroid surgery? Anesthesiology. 1991 Nov;75(5):918-9. doi: 10.1097/00000542-199111000-00036. No abstract available. PMID 1952223
- [Background] Greatorex RA, Denny NM. Application of the laryngeal mask airway to thyroid surgery and the preservation of the recurrent laryngeal nerve. Ann R Coll Surg Engl. 1991 Nov;73(6):352-4. PMID 1759763
- [Background] Akhtar TM. Laryngeal mask airway and visualisation of vocal cords during thyroid surgery. Can J Anaesth. 1991 Jan;38(1):140. doi: 10.1007/BF03009184. No abstract available. PMID 1989734
- [Derived] Kotsovolis G, Pliakos I, Panidis S, Gkinas D, Papavramidis T. Comparison Between the Protector Laryngeal Mask Airway and the Endotracheal Tube for Minimally Invasive Thyroid and Parathyroid Surgery. World J Surg. 2019 Nov;43(11):2822-2828. doi: 10.1007/s00268-019-05122-8. PMID 31410514